CLINICAL TRIAL: NCT00781690
Title: Pilot, Prospective, Multicenter, Open and Non-randomised Study: Definition of an Index of Anti Xa Value at the End of Hemodialysis Treatment.
Brief Title: Reduction of Heparin Dose in Dialysis With Evodial System
Acronym: RHODES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vantive Health LLC (Industry)
Collaborators: Gambro Lundia AB (Industry); Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1456; ISRCTN 93952087
Record Dates: First submitted 2008-10-28; First posted 2008-10-29 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Chronic Kidney Failure
Keywords: Chronic kidney failure; Heparin; Hemodialysis; Biocompatibility
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Treatment with Evodial with reduction of heparin across study period
  Interventions: Device: Evodial hemodialysers and Evodia blood lines

INTERVENTIONS:
Device: Evodial hemodialysers and Evodia blood lines — Maximum 8 weeks treatment with Evodial dialysers with reduction of heparin dose

SUMMARY:
The current clinical study aims at defining an index of Anti Xa, which is the marker to evaluate the activity of heparin, at the end of the dialysis treatment and so showing the possibility to decrease heparin doses during hemodialysis when using Evodial hemodialyzer. Actually, an elevated value of AntiXa at the end of the dialysis treatment increases the risk of bleeding for patients with diabetic retinopathy, or for instance in case of fall at home.

DETAILED DESCRIPTION:
In parallel to the new hemodialyzer, Evodia blood lines were developed to improve characteristics of the extracorporeal circuit in term of reduced activation of the coagulation system and lower deposits of clot components.

The aim is to provide a system (hemodialyzer and extracorporeal circuit) with a low thrombogenicity and that can be used with low heparin dose in order to reduce the patients' bleeding risk at the end of HD treatment.

Measurements of TAT (Thrombin-Antithrombin), the marker of the activation of the coagulation, will be performed during the study in order to evaluate the thrombogenicity of the system.

The ionic clearance will be collected during all treatments to evaluate the performance of the hemodialyzer.

The study will be divided into three steps

* Period 1: Usual heparin dose with usual hemodialyzer and standard blood lines (baseline),
* Period 2: Decrease of heparin dose with Evodial hemodialyzer and standard bloodlines
* Period 3: Lowest heparin dose defined in step 2 using the system Evodial hemodialyzer and SMA bloodlines.

Each patient included into the study will perform the three steps. As the risk of extracorporeal circuit clotting will be rather important, no control group (usual hemodialyzer with heparin decrease dose) will be performed.

ELIGIBILITY:
Inclusion criteria

* Patients suffering from chronic renal failure,
* Patients treated in HD three times a week for at least 3 months, with a stable heparin dose and the same filter,
* Patients treated in 4-4.5 hours HD mode with a blood flow between 300-350 ml/min,
* Patients for whom either LMWH (Enoxaparin, Nadroparin, Tinzaparin) or UFH is used,
* Patients with a well-functioning vascular access as judged by the investigator,
* Patients treated either on AK, Innova or Integra dialysis machines equipped with ionic dialysance device,
* Patients older than 18 years,
* Patients with negative serologies (AIDS, Hepatitis)
* Patients having signed consent to participate in the study.

Exclusion criteria

* Patient with HIT or known heparin allergy,
* Patient treated in HD in single needle mode,
* Patients with catheter,
* Patients with acute inflammatory event that may affect, as judged by investigator patients' safety or study results,
* Patients participating in other studies that could interfere with the objective of this study,
* Patients with active malignant disease,
* Patients receiving heparin outside dialysis treatment,
* Patients under guardianship,
* Pregnant women, nursing mothers and women planning a pregnancy during the course of this study,
* Patients with serious history of coagulopathy,
* Patients receiving Anti-Vitamin K medication,
* Patients receiving an association of anti platelets agents,
* Patients with heparin dose that can not be reduced for technical reason (excluding patients receiving too low heparin dose with no possibility of further reduction).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2008-09; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
The primary criterion is the measurement of Anti Xa at the end of dialysis sessions. | End of dialysis treatment

SECONDARY OUTCOMES:
Follow-up of aPTT for patients treated with UFH, | Kinetic on single dialysis treatment
Evaluation of TAT (Thrombin-Antithrombin) complex, | Kinetic on single dialysis treatment
Follow-up of ionic clearance (Diascan) measurements during HD sessions, | Kinetic of single dialysis treatment
Evaluation of the quality of the rinse-back (filter and circuit) via a visual scale, | End of dialysis treatment
Follow-up of AE/SAE. | All treatments during study period

CONTACTS AND LOCATIONS:
Overall Officials: Michèle Kessler, Pf, Study Chair — Hopital Brabois, Vandoeuvre les Nancy
Locations (7):
- France (4):
  - Calydial dialysis unit, Irigny
  - Clinique St Exupéry, Toulouse
  - Hopital Brabois, Vandœuvre-lès-Nancy
  - ALTIR Dialysis center, Vandœuvre-lès-Nancy
- Medizinische Hochschule, Hanover, Germany
- Borgo Trento Hospital, Verona, Italy
- Karolinska Hospital, Stockholm, Sweden

REFERENCES:
- [Background] Lavaud S, Canivet E, Wuillai A, Maheut H, Randoux C, Bonnet JM, Renaux JL, Chanard J. Optimal anticoagulation strategy in haemodialysis with heparin-coated polyacrylonitrile membrane. Nephrol Dial Transplant. 2003 Oct;18(10):2097-104. doi: 10.1093/ndt/gfg272. PMID 13679486
- [Background] Chanard J, Lavaud S, Maheut H, Kazes I, Vitry F, Rieu P. The clinical evaluation of low-dose heparin in haemodialysis: a prospective study using the heparin-coated AN69 ST membrane. Nephrol Dial Transplant. 2008 Jun;23(6):2003-9. doi: 10.1093/ndt/gfm888. Epub 2007 Dec 21. PMID 18156457
- [Derived] Kessler M, Gangemi C, Gutierrez Martones A, Lacombe JL, Krier-Coudert MJ, Galland R, Kielstein JT, Moureau F, Loughraieb N. Heparin-grafted dialysis membrane allows minimal systemic anticoagulation in regular hemodialysis patients: a prospective proof-of-concept study. Hemodial Int. 2013 Apr;17(2):282-93. doi: 10.1111/j.1542-4758.2012.00733.x. Epub 2012 Aug 23. PMID 22925178